CLINICAL TRIAL: NCT02682589
Title: A Multicenter, Prospective, Randomized Clinical Trial to Investigate Open Versus Laparoscopic Complete Mesocolic Excision for Locally Advanced Colon Cancer
Brief Title: Open Versus Laparoscopic Complete Mesocolic Excision for Locally Advanced Colon Cancer
Acronym: OLCMECC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: West China Hospital (Other); Changhai Hospital (Other); Chinese PLA General Hospital (Other); Peking Union Medical College Hospital (Other); Ruijin Hospital (Other); RenJi Hospital (Other); Shanghai Changzheng Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Fujian Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yueming Sun, Director of the Colorectal Surgery Department, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRSYM201602
Record Dates: First submitted 2016-02-04; First posted 2016-02-15 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Colon Cancer
Keywords: Complete Mesocolic Excision; locally advanced Colon Cancer; Laparoscopic
MeSH Terms: conditions — Colonic Neoplasms | interventions — Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open surgery (Active Comparator): Patients undergo open CME. A standard midline incision carefully protected is made through the abdominal wall and the abdominal cavity is explored. A colectomy with CME is performed with the removal of the afflicted colon and its accessory lymphovascular supply at their origins by resecting the colon and mesocolon in an intact envelope of visceral peritoneum and mesenteric fascia.
  Interventions: Procedure: Open surgery
- Laparoscopic surgery (Experimental): Patients undergo laparoscopic CME. A small infraumbilical incision is made through the abdominal skin and the abdominal cavity is insufflated with carbon dioxide to allow access and visualization. The abdominal cavity is explored. A colectomy with CME is performed using laparoscopic-assisted techniques. A 6-8cm midline auxiliary incision is made for specimen extraction and anastomosis.
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Open surgery — A traditional midline incision is made through the abdominal wall and a colectomy with CME is performed.
  Arms: Open surgery
Procedure: Laparoscopic surgery — 3-5 small incisions are made through the abdominal wall for the placement of trocars and the abdominal cavity is insufflated with carbon dioxide to allow access, visualization and operation. A 6-8cm auxiliary incision is made for specimen extraction and anastomosis. Conversion may occur due to technical difficulties or intraoperative complications, which is defined when completion of the dissection of the mesocolon is performed through a traditional open abdominal approach. Patients undergo conversion to laparotomy will be excluded from this study.
  Arms: Laparoscopic surgery

SUMMARY:
Randomized, multicenter, phase III trial to compare the short and long outcomes of laparoscopic CME with open CME in treating patients with locally advanced colon cancer.

DETAILED DESCRIPTION:
Laparoscopic complete mesocolic excision (CME) in treating colon cancer has been reported to be feasible and safe and holds many advantages when compared with traditional open surgery, such as reducing preoperative blood loss, alleviating postoperative pain and reducing complications and length of hospital stay. Whether laparoscopic CME could achieve an equivalent oncological outcome, especially for locally advanced malignancy, is still being discussed.

The purpose of this study is to determine the short and long outcomes of open and laparoscopic CME for locally advanced colon cancer patients. The primary endpoint is the 5-year disease-free survival rate. Secondary endpoints include completeness of mesocolon, morbidity and mortality, local recurrence, overall survival, quality of life et al.

In this study, eligible patient will be randomly allocated to receive either open or laparoscopic CME surgery. Randomization will be performed centrally and be stratified for age, gender, T-stage, tumor location. Patients will be randomized in a 2:1 ratio, in favor of the laparoscopic CME.

The extent of resection according to CME principle is identical for both arms. CME involves the removal of the afflicted colon and its accessory lymphvascular supply at their origins by resecting the colon and mesocolon in an intact envelope of visceral peritoneum and mesenteric fascia. Type of anastomosis, location of auxiliary incision and drainage of surgical field are up to the discretion of the surgeon. In laparoscopic surgery, a "medial-to-lateral" approach and a no-touch isolation are required .

Intraoperative pictures were taken at various stages, as were photographs of the postoperative specimen, which will be assessed by a third-party expert to qualify the surgery.

The baseline demographics and conditions as well as the perioperative and postoperative outcomes will be recorded through a prior designed format.

Our study is expected to last seven years, of which two years for recruiting patients, five years for follow-up. Patients are followed up every 3 months for 2 year, every 6 months for 3 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for curative surgery over 18 years old;
* American Society of Anesthesiologists(ASA) grade I-III;
* Pathological diagnosis of adenocarcinoma;
* Tumor located between the cecum and sigmoid colon;
* Enhanced CT scan of chest, abdominal and pelvic cavity: preoperative assessment of tumor stage is T3-T4 N0 or T any N+ (according to the National Comprehensive Cancer Network(NCCN) clinical practice guidelines in oncology: colon cancer version 2.2015);there is no distant metastasis;
* Informed consent;
* No preoperative chemoradiotherapy;
* No history of familial adenomatous polyposis, ulcerative colitis or Crohn's disease.

Exclusion Criteria:

* Pregnant patient;
* History of psychiatric disease;
* Use of systemic steroids;
* Conversion to laparotomy;
* Simultaneous or simultaneous multiple primary colorectal cancer;
* Preoperative imaging examination results show:

  1. Tumor involves the surrounding organs and combined organ resection need to be done;
  2. distant metastasis;
  3. unable to perform R0 resection;
* Postoperative pathology of T1-T2 N0;
* History of any other malignant tumor in recent 5 years;
* Patients need emergency operation: mechanic ileus, perforation.
* Not suitable for laparoscopic surgery (i.e., extensive adhesion caused by abdominal surgery, not suitable for artificial pneumoperitoneum, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2016-04; Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 5 years

SECONDARY OUTCOMES:
overall survival | 5 years
recurrence-free survival | 5 years
local recurrence rate | 5 years
length of postoperative hospital stay | 30 days
  Length of postoperative hospital stay is defined as a duration between surgery and first discharge. An expected average is 10 days.
early complication rate | 30 days
  Early complication is defined as a complication that occurred between the finish of the surgery and postoperative day 30. Complications includes anastomotic leakage, anastomotic bleeding, chyle leakage, wound infection, pulmonary embolism, myocardial infarction et al.The Clavien-Dindo Classification of Surgical Complications will be applied to access the degree of severity of postoperative complications.
operative time | 1 day
completeness of the mesocolon of the specimen | 1 day
  A central review by pathologists to define the completeness of the mesocolon to be good, moderate or poor will be performed on the specimen photographs.
number of lymph nodes retrieved | 1 day
postoperative quality of life as assessed by EORTC QLQ-C30 questionnaire | 5 years
  Compare the differences in postoperative quality of life of patients treated with these two regimens using EORTC QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fumin Zhang, Professor, Study Director — Ethics Committee of the First Affiliated Hospital, Nanjing Medical University, Jiangsu Province Hospital
Locations (1):
- Jiangsu province hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No